CLINICAL TRIAL: NCT03328780
Title: Prevalence of Anemia in Orthopedic Surgery, Data Collection From Classical Laboratory Determination of Hemoglobin, by Non-invasive Hemoglobin Measurement (Rad-67™) and by HemoCue®.
Brief Title: Anemia in Orthopedic Surgery - Determination of Hb
Status: Completed | Type: Observational
Sponsor: Theusinger Oliver M. (Other)
Responsible Party: Sponsor-Investigator, Theusinger Oliver M., Consultant, Priv. Doz. Dr. med., Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Other Study IDs: BASEC-Nr:2017-01361
Record Dates: First submitted 2017-10-26; First posted 2017-11-01 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Anemia
Keywords: preoperative; orthopedic surgery
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Hemoglobin determination: In this study classical laboratory determination, determination with HemoCue® and Rad-67™ will be performed to compare precision of those three methods as well as their correlation.
  Interventions: Device: Hemocue and Rad-67 measurement

INTERVENTIONS:
Device: Hemocue and Rad-67 measurement — Measurement of the hemoglobin level

SUMMARY:
Anemia prevalence in orthopedic surgery is up to 30 %. Identifying those patients prior to surgery and treating them would be ideal. Different ways of determining hemoglobin Levels are available. In this study classical laboratory determination, determination with HemoCue® and Rad-67™ will be performed to compare precision of those three methods as well as their correlation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Scheduled for elective orthopedic surgery
* Written informed consent.

Exclusion Criteria:

• Not able to speak the german language

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for elective orthopedic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Precision | through study completion, an average of 1 year
  Precision of the Masimo Rad-67 versus standard hemoglobin determination in the laboratory and the Hemocue (Correlation, Standard deviation, possible significant differences).

SECONDARY OUTCOMES:
Anemia | through study completion, an average of 1 year
  Prevalence of anemia in elective orthopedic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Oliver M Theusinger, MD, Study Director — Balgrist University Hospital
Locations (1):
- University Hopsital Balgrist, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No